CLINICAL TRIAL: NCT00764088
Title: A Retrospective Analysis of Patients With Full Thickness Wounds on a Case by Case Basis
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-008
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Full Thickness Wounds
Keywords: full Thickness wounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Anaysis of Full Thickness wounds: To demonstrate the effectiveness or ineffectiveness of novel treating agents or agents used for compassionate rescue, subjects and their wounds will be analyzed retrospectively and their non-identifiable information will be compiled in the form of case studies. Subjects who demonstrated characteristics of interest (e.g. healing) as determined by the PI will be chosen for case studies.

SUMMARY:
To demonstrate the effectiveness or ineffectiveness of novel treating agents or agents used for compassionate rescue, subjects and their wounds will be analyzed retrospectively and their non-identifiable information will be compiled in the form of case studies. Subjects who demonstrated characteristics of interest (e.g. healing) as determined by the PI will be chosen for case studies.

DETAILED DESCRIPTION:
All wounds at the Southwest Regional Wound Care Center (WCC) are managed using anti-biofilm strategies. When determining the therapeutic course for a patient and his full thickness wound, all management agents that are available are considered for use; and the clinician uses his judgment to determine the most appropriate tools to use that will give the patient the most likely chance of success. Some of the agents that are used are novel, and it is appropriate to demonstrate to others the potential usefulness of these agents

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years old
* Retrospective analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic- Southwest Regional Wound Care Center
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Retrospective Analysis of Patients with Full Thickness Wounds | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center